CLINICAL TRIAL: NCT01962727
Title: Scapular Dyskinesis: a Reliability and Validity Study of Comprehensive Classification Test
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201112034RIB
Record Dates: First submitted 2013-08-12; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Unilateral Shoulder Pain With and Without Scapular Dyskinesis
Keywords: scapular dyskinesis, kinematics, muscular activities

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study Design: Clinical measurement (cross-sectional)

Objectives: The purpose of this study was to investigate the reliability and validity of the novel scapular dyskinesis classification test.

Background: A visual-based clinical assessment with sufficient reliability and validity to identify scapular dyskinesis provides information for rehabilitation treatment.

Methods: A visual-based palpation method was evaluated by two independent physiotherapists in 60 subjects with unilateral shoulder pain to test reliability. This method classified the scapular movements during arm raising/lowing movements in scapular plane as single abnormal scapular patterns (inferior angle/ medial border/ superior border of scapula prominence and abnormal scapulohumeral rhythm) or mixed abnormal scapular patterns. Different patterns of scapular dyskinesis were also validated by corresponding alternation of the scapular kinematics and muscular activities assessed by electromagnetic motion-capturing system and surface electromyography (EMG).

DETAILED DESCRIPTION:
No other detailed description

ELIGIBILITY:
Inclusion Criteria:

* (1) they were from 18 to 50 years old and (2) they had unilateral shoulder pain around shoulder complex during activities.

Exclusion Criteria:

* history of shoulder dislocation, fracture, or shoulder surgery within past 1 year, or a history of direct contact injury to the neck if upper extremities within the past 1 month, scoliosis or excessive kyphosis, neurological disorders, body mass index (BMI)≧25, or demonstrate pain (VAS>3) during overall testing procedure.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sixty subjects (36 males and 14 females, age: 22.5 ± 2.6) were recruited.Potential participants from outpatient clinic in a University hospital and local internet media were evaluated and recruited. They read and signed the informed consent approved by the Hospital institutional review boards.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Reliability of scapular dyskinesis test | 2 hours
  The inter-rater reliability for the comprehensive scapular dyskinesis classification test was described using percentage of agreement and κ coefficient.
  Rating of scapular dyskinesis was evaluated and classified into 8 patterns including(A) patterns I (B) patterns II (C) pattern III (D) pattern IV (E) pattern I+II (F) pattern II+III (G) pattern I+III (H) pattern I+II+III.

SECONDARY OUTCOMES:
Validity of scapular dyskinesis test | 2 hours
  Different patterns of scapular dyskinesis were validated by corresponding alternation of the scapular kinematics and muscular activities assessed by electromagnetic motion-capturing system and surface electromyography.
  To quantitatively characterize the scapular kinematics and muscular activities, the kinematic data at 30°, 60°, 90°, and 120° and EMG data at 0~30°, 30°~60°, 60°~90°, 90°~120°, and >120° in the raising and lowering phases of humeral movement in the scapular plane were used as dependent variables. Data from the same scapular dyskinesis pattern assessed by 2 raters were used for validity analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jiu-Jenq Lin, PhD, Principal Investigator — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, 100 Taipei, Taiwan
Locations (1):
- Performance analysis laboratory, Taipei, Taiwan

REFERENCES:
- [Derived] Huang TS, Ou HL, Huang CY, Lin JJ. Specific kinematics and associated muscle activation in individuals with scapular dyskinesis. J Shoulder Elbow Surg. 2015 Aug;24(8):1227-34. doi: 10.1016/j.jse.2014.12.022. Epub 2015 Feb 19. PMID 25704212